CLINICAL TRIAL: NCT01833299
Title: Transcatheter Arterial Chemoembolization Combined With Sorafenib for Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TACE-Sorafenib
Record Dates: First submitted 2011-04-13; First posted 2013-04-16 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hepatocellular Carcinoma; Face Cancer
Keywords: TACE; Sorafenib; overall survival; time to progression
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the radiologists who assessed the outcomes were blinded.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE group (Active Comparator): Transcatheter arterial chemoembolization drugs and dosage:TACE with chemothrapy drugs (E-ADM 50mg, carboplatin 300 mg, MMC 8mg)and followed with embolization with lipiodol and absorbable gelatin sponge particles or polyvinyl alcohol particles.
  Interventions: Procedure: TACE
- TACE+sorafinib (Experimental): TACE+sorafinib
  Interventions: Procedure: TACE-Sorafenib group

INTERVENTIONS:
Procedure: TACE-Sorafenib group — Transcatheter arterial chemoembolization drugs and dosage:TACE with chemothrapy drugs (E-ADM 50mg, carboplatin 300 mg, MMC 8mg)and followed with embolization with lipiodol and absorbable gelatin sponge particles or polyvinyl alcohol particles.
  Oral sorafenib (400 mg BID) will be start the 2-4 weeks after the first TACE treatment and will continue until the patient shows disease progression, until unacceptable toxicity occurs, or until study termination.
  Other Names: TACE combined with Sorafenib
  Arms: TACE+sorafinib
Procedure: TACE
  Arms: TACE group

SUMMARY:
Hepatocellular carcinoma (HCC) is the 6th most common cancer and the third most frequent cause of cancer death worldwide. Hepatic resection (HR) has been the standard treatment modality for HCC aiming at clinical cure. In both Europe and Unit States proposed guidelines for HCC, HR was recommend only for patients with a single HCC lesion and preserved liver function . Unfortunately, only 10%-30% of HCCs are amenable to such "curative" surgical resection at the time of diagnosis, because of tumor multifocality, portal vein invasion, and underlying advanced liver cirrhosis . Alternatively, transarterial chemoembolization (TACE) has become the most popular modality for palliative treatment for the other patients. However, the long term outcomes were generally poor for HCC patients treated with TACE.

Recently, sorafenib has shown some promises in improvement of 3-month survival among patients with advanced HCC. It is claimed that sorafenib has become the standard of care for patients advanced HCC.

Thus, the purpose of this study was to prospectively compare the effectiveness of sorafenib combined with TACE with that of TACE alone in the treatment of unresectable HCC .

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common cause of cancer mortality in Asia. Most patients present with intermediate or advanced disease. Percutaneous ethanol injection, radiofrequency ablation, and transcatheter arterial chemoembolization (TACE) are not considered as a curative treatment and have achieved very limited success in eradicating large HCC.

Two phase III trials were shown to be efficacious and well-tolerated in patients with advanced HCC. Median overall survival was significantly 2 to 3 months longer in the sorafenib group than that in the placebo. It is interesting to recognize the combined therapeutic effect of TACE with sorafenib. The proposed study will make an important contribution to understanding not only the safety and efficacy of sorafenib in addition to TACE in patients diagnosed with unresectable HCC, but this will also be the first clinical trial prospectively to compare the effectiveness of sorafenib combined with TACE with that of TACE alone in the treatment of unresectable HCC

ELIGIBILITY:
Inclusion Criteria:

1. Adults patients ( 18-75 years of age) with a diagnosis of HCC which is not amenable to surgical resection or local ablative therapy
2. Histological confirmed HCC or clinical/laboratory diagnosis of HCC or nodules larger than 2 cm with typical vascular features or AFP > 200
3. Patient must have quantifiable disease limited to the liver
4. Patients must have at least one tumor lesion that meets both of the following criteria:
5. The lesion can be accurately measured in at least one dimension according to RECIST criteria
6. The lesion has not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
7. ECOG performance status (PS) <2
8. No prior targeted antiangiogenic therapy. Metronomic chemotherapies are allowed. At least 4 weeks since prior systemic chemotherapy,At least 4 weeks since prior TACE, At least 4 weeks since prior interferon.
9. Not pregnant
10. No significant baseline liver dysfunction. Cirrhotic status of Child-Pugh class A only
11. No significant renal impairment (creatinine clearance < 30 mL/minute) or patients on dialysis
12. No current infections requiring antibiotic therapy
13. Not on anticoagulation or suffering from a known bleeding disorder
14. No unstable coronary artery disease or recent MI

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from HCC except cervical carcinoma in situ, treated basal-cell carcinoma of the skin, superficial bladder tumors (Ta, Tis & T1), and any cancer curatively treated > 3 years prior to entry is permitted
2. Renal failure requiring hemo- or peritoneal dialysis
3. Child-Pugh B & C hepatic impairment
4. History of cardiac disease: > NY Heart Association (NYHA) class 2 congestive heart failure, active coronary artery disease, cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, and uncontrolled hypertension. Myocardial infarction more than 6 months prior to study entry is permitted.
5. Active clinically serious infections (> CTCAEv3 grade 2)
6. Known history of HIV
7. Known central nervous system tumors including metastatic brain disease
8. History of organ allograft
9. Substance abuse (current), psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
10. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
11. Patients unable to swallow oral medications.
12. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of the study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
13. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
14. Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg, despite optimal medical management
15. Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
16. Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug
17. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
18. Serious non-healing wound, ulcer, or bone fracture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of sorafenib combined with TACE | 1 year
  Measure:overall survival Measured from the date of TACE until the date of death or last visit

SECONDARY OUTCOMES:
Time to progression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: min-shan chen, M.D. Ph.D., Principal Investigator — Department of Hepatobiliary Surgery, Cancer Centre of Sun Yat-Sen University
Locations (1):
- Cancer Centre of Sun Yat-Sen University, Guangzhou, China

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin 2005;55:74-108. Llovet JM, Real MI, Montan˜a X, et al. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002;359:1734-59. Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, et al. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008;359:378-90. Bruix J, Llovet JM. Major achievements in hepatocellular carcinoma. Lancet 2009 21;373:614-616.